CLINICAL TRIAL: NCT05544409
Title: Early Implementation of MAKv1 Exoskeleton in TKA Rehabilitation
Brief Title: MAKv1 Exoskeleton for TKA Patients: a Safety, Usability and Clinical Effects Trial of an Early Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TKA_MAK
Record Dates: First submitted 2022-09-12; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Total Knee Arthroplasty
Keywords: exoskeleton; total knee arthroplasty; rehabilitation; MAKv1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAKv1 (Experimental): The MAKv1 group will receive 1 hour of MAKv1 rehabilitation, thrice per week during 1 month
  Interventions: Device: MAKv1

INTERVENTIONS:
Device: MAKv1 — 1 hour sessions with the MAKv1 exoskeleton, thrice per week during 1 month

SUMMARY:
The present study analyzes the effects of using a portable single limb exoskeleton (MAKv1) in patients with total knee artrhoplasty (TKA). Safety, usability and clinical effects of an early intervention program with the device with an early implementation are studied.

DETAILED DESCRIPTION:
The present study will analyze the safety, usability and clinical effects of using the MAKv1 exoskeleton in TKA patients. The intervention will consist of 1 hour sessions with the MAKv1 device, thrice per week during 1 month. Safety measurements (serious adverse events, vitals, and auto-perceived pain) will be collected at each session with the device, along with the repetitions performed at each exercise assisted with the device. After the first week is completed, measurements regarding clinical effect will be collected. Also, at the end of the month were the participants receive the sessions with the device, clinical effects will be measured again, along with a questionnaire to collect the users' perception of the device (QUEST 2.0).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing TKA surgery

Exclusion Criteria:

* inability to understand simple instructions
* postoperative complications that may be a risk to use the exoskeleton
* other conditions that prevented mobilisation in early stages after TKA
* weight > 100 kg
* size < 150 cm
* size > 190 cm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | Through study completion, an average of 2 months
  event that causes death, life-threat, hospitalization, disability, congenital anomaly, or that requires intervention to prevent permanent impairment or damage

SECONDARY OUTCOMES:
Auto-perceived Pain | Through completion of the use of the device, during 1 month
  Presence of pain collected with VAS scale (0 to 10)
Heart Rate | Through completion of the use of the device, during 1 month
  Differences in heart rate beofre and after the use of the device (measured in beats/min)
Blood pressure | Through completion of the use of the device, during 1 month
  Differences in blood pressure before and after the use of the device (measured in mmHg)
Oxygen Saturation | Through completion of the use of the device, during 1 month
  Differences in oxygen satruation before and after the use of the device (measured in %SpO2)
Body Termperature | Through completion of the use of the device, during 1 month
  Differences in body temperature before and after the use of the device (measured in celsius)
Repetitions per exercise | Through completion of the use of the device, during 1 month
  The number of repetitions per exercise assissted by the MAKv1 device was recorded (mesaured in number of repetitions)
QUEST 2.0 scale | At the first month of the participation in the trial
  QUEST 2.0 scale is a usability scale which rates the perception of the user about the device.
Range of Motion at the knee | Mesaured at the first week, at the first month and at the second month (follow-up) from participation
  Range of motion of the knee, measured in degrees (º).
Muscle strength at the knee | Mesaured at the first week, at the first month and at the second month (follow-up) from participation
  Muscle strength of knee muscles, measured by the modified Medical Research Council scale (mMRC).
Knee circumference | Mesaured at the first week, at the first month and at the second month (follow-up) from participation
  Circumference of the knee, measured with a metric tape placed at the upper border of the patella (measured in cm)
Quadriceps circumference | Mesaured at the first week, at the first month and at the second month (follow-up) from participation
  Circumference of the quadriceps, measured with a metric tape placed at 10 cm from the upper border of the patella (measured in cm)
6MWT | Mesaured at the first month and at the second month (follow-up) from participation
  6MWT consists of a test were the subject is asked to walk for 6 minutes and the distance covered is collected (measured in meters)
TUG | Mesaured at the first month and at the second month (follow-up) from participation
  The Timed Up and Go test consists of a test were the subject is asked to stand up from a chair, cover 3 meters in a straight line, and then go back to sit in the same chair. Time to complete the task is recorded (measured in seconds)
FAC | Mesaured at the first month and at the second month (follow-up) from participation
  The functional Ambulation Categories scale measures the patient's ability according to the assistance needed to deambulate. A score is given from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Luisa López Morón, Principal Investigator — Hospital Universitario Sanitas La Zarzuela
Locations (1):
- Hozpital Universitario La Zarzuela, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be anonymized in order to avoid pariticpant's identification